CLINICAL TRIAL: NCT03622476
Title: Capital Characteristic Application: Pharmacokinetic（PK） Research on Chinese Children of Hemophilia
Brief Title: Pharmacokinetic (PK)Research on Chinese Children of Hemophilia
Acronym: PK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Runhui WU, Capital Medical Univercity, Beijing Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-PK-20180630
Record Dates: First submitted 2018-07-30; First posted 2018-08-09 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pharmacokinetics
Keywords: Hemophilia A，pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PK research (Experimental): Interventional studies were performed in the 1-7 year old subgroup, and the children received a comprehensive assessment and PK test every 3 months. After the 72-hour washout period, 50 IU/kg of concentrated FVIII was administered in a single dose, and blood was taken within half an hour before the infusion and 1 h, 9 h, 24 h, and 48 h after the infusion, and the samples were centrifuged. If the assessment considers that the treatment is inadequate, then the valley concentration target is upgraded.
  Interventions: Drug: concentrated FVIII

INTERVENTIONS:
Drug: concentrated FVIII — Intervention if the assessment considers that the treatment is inadequate

SUMMARY:
The study start on June 30, 2018. The Severe(F Ⅷ<1%) hemophilia A children without F Ⅷ inhibitor combining were recruited to Test the concentration of the drug in the blood to provide better treatment.

DETAILED DESCRIPTION:
Through the integration of two technologies, pharmacokinetics and comprehensive evaluation system, we can improve the individualized prevention and treatment of hemophilia in Chinese children and achieve precise customization of treatment plans. Rational use of medical resources, but also fully achieve the prevention and treatment goals.

ELIGIBILITY:
Inclusion Criteria:

* FⅧ<1% ,
* 1-14years old,
* There have been at least one history of bleeding in any joint of the knee, elbow, or ankle.
* A blood product containing FVIII is applied.
* There were no inhibitors at the time of enrollment, and there was no inhibitor-positive history and family history.
* Clinical visits are available on a regular basis and data is available, and preventive treatment is available prior to enrollment.
* The child was enrolled in the group and the guardian agreed.

Exclusion Criteria:

* Combining other disease researchers believes that it is not suitable for enrollment.
* FVIII inhibitor was found.
* Refuse to participate in research

Ages: 1 Year to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Estimated)
Dates: Start 2018-06-30 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasound evaluation | 3 years
  the sonographer will use ultrasound to assess whether the patient's joint lesions become more severe than when they were enrolled.
Imaging evaluation | 3 years
  the imaging specialist will use MRI to assess whether the patient's joint lesions are more severe than when they were enrolled.

SECONDARY OUTCOMES:
Annualized Bleeding Rate | 3 years
  How many times for all types of bleeding
Annualized Joint Bleeding Rate | 3 years
  How many times for joint bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No